CLINICAL TRIAL: NCT04304300
Title: Radiotherapy in IDH Mutated Glioma: Evaluation of Late Outcomes
Acronym: RIGEL
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: HollandPTC (Industry); Amsterdam University Medical Center (Other); Leiden University Medical Center (Other); Delft University of Technology (Other); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, Alejandra Mendez Romero, MD, PhD, Erasmus Medical Center
Other Study IDs: NL69780.078.19; Netherlands Trial Register (Registry Identifier: NL7993)
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Astrocytoma, Grade II; Astrocytoma, Grade III; Oligodendroglioma; Oligodendroglioma, Anaplastic
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, optional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Glioma, IDH mutated, grade 2 and 3

SUMMARY:
Rationale: Standard postoperative treatment of isocitrate dehydrogenase 1/2 mutated grade 2 and 3 glioma (IDHmG) consists of radiotherapy and chemotherapy. The improving prognosis of these patients leads towards more emphasis on the long-term effects of treatment. Specifically radiotherapy has been implicated in the development of delayed neurocognitive deterioration. The impact of modern radiotherapy techniques (such as intensity modulated radiotherapy, volumetric modulated radiotherapy and proton beam therapy) and chemotherapy on general toxicity, late neurocognitive outcomes and imaging changes is currently unclear.

Objectives:

* To report treatment outcomes and radiation-induced toxicity from a prospective, multicentre observational cohort of IDHmG patients treated with radiotherapy and chemotherapy,
* To integrate radiotherapeutic dose distributions, imaging changes and neuropsychological outcome in IDHmG.
* To evaluate the Dutch selection criteria for proton therapy applied to IDHmG based on the outcomes collected in this observational study.
* To assess the impact of proton and photon therapy on health-related quality of life (HRQoL) and health-related economics (HR-E) in IDHmG patients.
* To collect genetic material for future translational research into the interaction between germline DNA, prognosis and radiation-induced toxicity.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This project is a multicentre, observational cohort of patients undergoing radiotherapy and chemotherapy for IDHmG. The protocol closely follows the local guidelines for clinical follow-up. Specific to the study are extra questionnaires and specific imaging acquired during scheduled MRI's. Routine neuropsychological investigation is standard of care in Erasmus Medical Center (Erasmus MC), but not in all participating centers. We feel the additional burden of participation in this study to be low.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioma, World Health Organisation (WHO) grade 2 or 3, IDH mutated
* Indication for standard treatment with radiotherapy and chemotherapy. For WHO grade 2 tumors 50.4 Gy relative biological equivalent (RBE) in 28 fractions. For WHO grade 3 tumors 59.4 Gy (RBE) in 33 fractions.
* Ability to comply with the protocol, including neuropsychological testing and imaging.
* Ability to understand the requirements of the study and to give written informed consent, as determined by the treating physician.
* Written informed consent.

Exclusion Criteria:

* Any prior chemotherapy for IDHmG. This includes upfront postoperative chemotherapy.
* Any prior cranial radiotherapy, including but not limited to radiotherapy for IDHmG.
* Prior invasive malignancy, except non-melanoma skin cancer, completely resected cervical or prostate cancer (with current prostate specific antigen (PSA) of less than or equal to 0.1 ng/mL).
* Extensive white matter disease visible on pre-therapy imaging (Fazekas grade ≥2)
* Contra-indication for magnetic resonance (MR) imaging (i.e. metal implants, claustrophobia)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule in the participating hospitals
* Any other serious medical condition that could interfere with follow-up.
* Severe aphasia or language barrier interfering with assessing endpoints (i.e. completion of questionnaires or neurocognitive performance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IDH mutated glioma patients, WHO grade 2 and 3, who undergo postoperative radiotherapy and chemotherapy as standard treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Toxicity (selected CTCAE 5.0 items) | 24 months
  The Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 displays Grade 1 to 5, ranging from 'mild' to 'death'. The case report form will include a predefined set of CTCAE items of expected radiotherapy related toxicities. In addition, other CTCAE toxicities grade ≥ 2 that are likely, possibly or definitely related to the radiotherapy should be recorded in the case report form (CRF), when they occur. All items will include a causality assessment: likely or definitely attributable to radiotherapy, unrelated or unlikely attributable to radiotherapy, or not assessable.
Neurocognitive testing | 24 months
  Neurocognitive functioning will be assessed with a standard and well established short neuropsychological test battery, developed for use in clinical trials. The following tests are included: Hopkins Verbal Learning Test (HVLT), Trail Making Test part A and B (TMT A/B), Controlled Oral Word Association (COWA), Medical Outcomes Study Cognitive Functioning Scale (MOS), Diagnostic Instrument for Mild Aphasia (DIMA)

SECONDARY OUTCOMES:
Next intervention free survival (NIFS) | 48 months
  NIFS is defined as time from first irradiation to date of initiation of further treatment after radio- and/or chemotherapy or death (any cause), whichever occurs first.
Progression Free Survival (PFS) | 48 months
  PFS is defined as the time from first irradiation to progressive disease, according to (any of) the Response Asessment in Neuro Oncology (RANO) criteria for progressive disease in low grade glioma.
Overall Survival (OS) | 48 months
  OS is defined as time from first irradiation to date of death from any cause.
Health Related Quality of Life (HRQOL) | 24 months
  HRQoL will be assessed with the EORTC quality of life questionnaire (QLQ-C30) supplemented by the neuro-oncological module (QLQ-BN20) and the Euro Quality of Life questionnaire (EQ5D-5L)
Health - Related Economics | 24 months
  For the Health Related Economics (HR-E) analyses, the EQ5D - 5L questionnaire will be used in conjunction with the Productivity Costs Questionnaire (iPCQ) and the Medical Consumption Questionnaire (iMCQ). These questionaires are optional.

OTHER OUTCOMES:
Radiological data | 4 months
  If feasible, pre- and 4 months post-treatment a scan protocol will be used that, besides the standard clinical imaging, will focus on (micro-)structural and microvascular characteristics that could predict neurocognitive outcome and treatment efficacy. This feasibility is site-specific.

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Erasmus MC, Rotterdam, South Holland
  - Amsterdam UMC, Amsterdam
  - HollandPTC, Delft
  - Leiden University Medical Center, Leiden
  - Haaglanden Medical Center, Leidschendam

IPD SHARING:
Plan to Share IPD: No